CLINICAL TRIAL: NCT00005841
Title: A Phase I Trial of a Vaccine Combining Tyrosinase/GP100/Mart-1 Peptides Emulsified With Montanide ISA 51 With ProGP for Patients With Resected Stages III and IV Melanoma
Brief Title: Vaccine Therapy in Treating Patients With Stage III or Stage IV Melanoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Toxicity/Side Effects
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000067857 (10M-99-3); LAC-USC-10M993; LAC-USC-IRB-99B028; NCI-470
Record Dates: First submitted 2000-06-02; First posted 2004-05-26 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Intraocular Melanoma; Melanoma (Skin)
Keywords: iris melanoma; ciliary body and choroid melanoma, small size; ciliary body and choroid melanoma, medium/large size; extraocular extension melanoma; recurrent intraocular melanoma; stage III melanoma; stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Uveal Melanoma; Melanoma | interventions — MART-1 Antigen; incomplete Freund's adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: MART-1 antigen
Biological: gp100 antigen
Biological: incomplete Freund's adjuvant
Biological: progenipoietin
Biological: tyrosinase peptide

SUMMARY:
RATIONALE: Vaccines made from melanoma cells may make the body build an immune response to kill tumor cells. Vaccine therapy plus filgrastim combined with a specific protein may be a more effective treatment for melanoma.

PURPOSE: This phase I trial is studying the side effects and best dose of vaccine therapy in treating patients with stage III or stage IV melanoma that has been completely removed during surgery.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of filgrastim (G-CSF)-fetal liver tyrosine kinase-3 (Flt3K) fusion protein when combined with melanoma peptide vaccine comprising tyrosinase:368-376 peptide, gp100:209-217 antigen, and MART-1:26-35 antigen emulsified in Montanide ISA-51 in patients with completely resected stage III or IV melanoma. II. Determine the toxicity and safety of this regimen in these patients. III. Determine the immune responses to tyrosinase, MART-1, and gp100 antigens in patients before, during, and after receiving these vaccinations.

OUTLINE: This is a dose escalation, multicenter study of filgrastim (G-CSF)-fetal liver tyrosine kinase-3 (Flt3K) (G-CSF-Flt3K) fusion protein. Patients receive melanoma peptide vaccine comprising tyrosinase:368-376 peptide, gp100:209-217 antigen, and MART-1:26-35 antigen emulsified in Montanide ISA-51 subcutaneously (SQ) monthly for 6 months, and then at 9 and 12 months for a total of 8 vaccinations. Patients receive G-CSF-Flt3K fusion protein SQ daily for 3 days before, immediately after, and then daily for 6 days after each vaccination. Cohorts of 6-10 patients receive escalating doses of G-CSF-Flt3K fusion protein until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6-10 patients experience dose limiting toxicity. Patients are followed every 3 months through year 2 after resection, every 6 months for 3 years, and then annually thereafter until disease progression.

PROJECTED ACCRUAL: A total of 30-50 patients will be accrued for this study within 12-18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven completely resected stage III or IV cutaneous, mucosal, or ocular melanoma Disease free, but at high risk of relapse Must meet 1 of the following criteria: Failed interferon alfa (IFN-A) therapy Ineligible for IFN-A therapy Refused IFN-A therapy HLA-A2.1 positive Availability of tumor tissue for analysis of gp100 antigen staining with antibody HMB-45, and for expression of tyrosinase and MART-1 antigens by immunohistochemistry Tumor cells must be positive for at least 1 antigen

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0 or 1 Life expectancy: Not specified Hematopoietic: WBC at least 3,000/mm3 Granulocyte count at least 1,500/mm3 Hemoglobin at least 9.0 g/dL Platelet count at least 100,000/mm3 No coagulation or bleeding disorders Hepatic: Bilirubin no greater than 2.0 mg/dL SGOT and SGPT no greater than 2.5 times upper limit of normal Renal: Creatinine no greater than 2.0 mg/dL Cardiovascular: No concurrent major medical illness of the cardiovascular system Pulmonary: No concurrent major medical illness of the respiratory system Immunologic: Hepatitis B surface antigen negative and hepatitis C antibody negative HIV negative No history of uveitis or other autoimmune inflammatory eye disease No other active autoimmune disease No known allergic reaction to Montanide ISA-51 Other: No concurrent major systemic infection including pneumonia or sepsis No concurrent major medical illness of the gastrointestinal system Not pregnant or nursing Negative pregnancy test No other malignancy within the past 5 years except curatively treated squamous cell skin cancer or carcinoma in situ of the cervix allowed 30 days after treatment

PRIOR CONCURRENT THERAPY: Biologic therapy: See Disease Characteristics No prior tyrosinase:368-376 peptide, gp100:209-217 antigen, or MART-1:26-35 antigen Chemotherapy: Not specified Endocrine therapy: No concurrent steroids Radiotherapy: At least 1 month since prior radiotherapy No concurrent radiotherapy Surgery: See Disease Characteristics Other: At least 1 month since other prior therapy, including adjuvant therapy, for melanoma No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2000-06; Primary Completion 2000-12 (Actual); Study Completion 2002-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey S. Weber, MD, PhD, Study Chair — University of Southern California
Locations (2):
- United States (2):
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - City of Hope National Medical Center, Los Angeles, California

REFERENCES:
- [Result] Pullarkat V, Lee PP, Scotland R, Rubio V, Groshen S, Gee C, Lau R, Snively J, Sian S, Woulfe SL, Wolfe RA, Weber JS. A phase I trial of SD-9427 (progenipoietin) with a multipeptide vaccine for resected metastatic melanoma. Clin Cancer Res. 2003 Apr;9(4):1301-12. PMID 12684398